CLINICAL TRIAL: NCT03998722
Title: An Open Single-arm Investigation to Evaluate the Use of VagiVital® for Treatment of Vaginal Atrophy in Cancer Patients Undergoing Adjuvant Aromatase Inhibitor Therapy - 12 Weeks Follow-up
Brief Title: Evaluation of VagiVital® for Treatment of Vaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vagipep101
Record Dates: First submitted 2019-05-24; First posted 2019-06-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Intervention Model Description: An open single-armed study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vagivital (Experimental): Vagivital once Daily for 12 weeks
  Interventions: Device: Vagivital

INTERVENTIONS:
Device: Vagivital — Vagivital once Daily for 12 weeks

SUMMARY:
An open study to evaluate the ability of VagiVital in reducing the severity of moderate to severe symptoms of vaginal atrophy for women under treatment on adjuvant aromatase inhibitor therapy. Vaginal pH and a self-assessment of the symptoms will be assessed. The treatment consists of administration of intravaginal gel from an applicator filled from a tube, once daily for 12 weeks. All participants will self- administer the intravaginal gel once daily for 12 weeks.

DETAILED DESCRIPTION:
Management of breast cancer involves systematic therapies including chemotherapy and endocrine therapy which can lead to vaginal atrophy (VA), caused by decreased levels of circulating estrogen to urinary and vaginal receptors. Due to the reduced estrogen production, less vaginal fluid is produced within the vagina and the mucosa becomes thinner and more fragile. This group of patients can not use estrogen treatment to reduce the symptoms of vaginal atrophy.

A previous study showed a significant reduction in the severity of the most bothersome VA symptoms and vaginal pH was improved (decreased) as well as increased percentage of superficial cells over a 12 week treatment period with Vagivital.

In this study all participants will self- administer the intravaginal gel once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

To participate in the investigation, a subject must:

1. Be a female, 18 years or older, who is willing to participate in the study as indicated by signing the informed consent.
2. Women over the age of 18 who have been diagnosed with cancer and are currently taking adjuvant AI therapy who also complain of vaginal atrophy symptoms including vaginal dryness, vaginal itching, frequent urinary tract infections, or dyspareunia are candidates for this study. They also have to be sexually active or wanted to be so, but couldn´t because of problems with vaginal atrophy.
3. Have one moderate to severe VA symptom (vaginal irritation and itching, vaginal dryness, dysuria, dyspareunia or presence of vaginal bleeding associated with sexual activity) that has been identified by the subject as being the most bothersome to her according to the scale presented in APPENDIX B.
4. Be judged by the Principal Investigator as being in otherwise good health based on the medical evaluation performed at baseline. The medical evaluation findings must include:

   1. A normal or clinically non-significant finding at physical examination, including vital signs (blood pressure and heart rate).
   2. A normal or clinically non-significant finding at gynecological examination.
   3. A normal or clinically non-significant finding at clinical breast examination. An acceptable breast examination is defined as an examination in which no masses or other findings are identified which are suspected of being malignant.
   4. Urine analysis test results within reference limits or with non-significant deviations from reference values.
   5. A sitting systolic blood pressure ≤ 150 mmHg and diastolic blood pressure ≤ 90 mmHg at screening. Hypertensive subjects controlled with stable medications, who have a blood pressure ≤ 150 (systolic) and ≤ 90 (diastolic) mmHg are suitable for inclusion
5. Be willing to abstain from sexual activity and the use of vaginal douching within 24 hours prior to vaginal pH measurements at screening and at Visits 2 and 3.

Exclusion Criteria:

To participate in the investigation, a subject must not:

1. Be currently hospitalized.
2. Have a history of ongoing cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or Sub-Investigator.
3. Have a history of undiagnosed vaginal bleeding.
4. Have an ongoing urogenital infection at the screening visit.
5. Any contraindication to the gel (VagiVital) therapy and allergy to the use of any components of the investigational device.
6. Have a history of drug and/or alcohol abuse within one year of start of study.
7. Have used any prescription or OTC medications including phytoestrogens, herbal medicinal products or hormonal intra-uterine device with known estrogenic effects within 12 weeks prior to screening procedures.
8. Have used any type of vaginal lubricants and moisturizers within 24 hours prior to screening procedures.
9. Have used estrogen alone or estrogen/progestin for any of the following time periods:

   1. Vaginal hormonal products (rings, creams, gels, vaginal suppositories) within 12 weeks prior to Screening procedures;
   2. Transdermal estrogen alone or estrogen/progestin products including percutaneous estrogen gels for at least 12 weeks prior to screening procedures.
   3. Oral estrogen and/or progestin therapy within 12 weeks prior to Screening procedures;
   4. Intrauterine progestin therapy within 12 weeks prior to Screening procedures;
   5. Progestin implants and estrogen alone injectable drug therapy within 12 weeks prior to screening procedures;
   6. Estrogen pellet therapy or progestational injectable drug therapy within 6 months prior to screening procedures;
10. Have any reason, which in the opinion of the Principal Investigator would prevent the subject from safely participating in the study or complying with protocol requirements.
11. Have participated in another clinical trial within 90 days prior to screening, have received an investigational drug within the three months prior to the initial dose of study medication, or be likely to participate in another clinical trial or receive another investigational medication during the study.
12. Have contraindication to any planned study procedure.
13. Fulfils any other reason for exclusion as stated by the Declaration of Helsinki.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Change in severity of VA symptom | 12 weeks
  Change from baseline to Week 12 in severity of VA symptom (vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or presence of vaginal bleeding associated with sexual activity) that has been self-identified by the subject as being the most bothersome to her.The VA Symptoms are graded from 0-3, where 0 = none and 3 = severe

SECONDARY OUTCOMES:
Change in Vaginal pH | 4 weeks
  Change from baseline to Week 4 in Vaginal pH
Change in Vaginal pH | 12 weeks
  Change from baseline to Week 12 in Vaginal pH
Change in severity of VA Symptom | 4 weeks
  Change from baseline to Week 4 in severity of the VA symptoms (vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or presence of vaginal bleeding associated with sexual activity). The VA Symptoms are graded from 0-3, where 0 = none and 3 = severe
Change in total score in Quality of Life evaluation parameters | 12 weeks
  Change from baseline to Week 12 in Quality of Life evaluation parameters Women's Health Questionnaire. Total Score (sum of the questions as recorded in the data management system (Yes, definitely=0, Yes, sometimes=1, No, not much=2 or No, not at all=3) except for question 7, 8, 10, 12 and 14 where the score opposite in points. Missing values are imputed using the mean of all recorded values. Analysis set ITT.
Number of AEs and assessment of intensity, causality and seriousness of Advers Events | 14 weeks
  The adverse events will be classified as non-serious adverse event or serious adverse event (SAE), the intensity will be graded as mild, moderate or severe and causality will be classified as unlikely, possible and probably.
Change in Blod pressure | 4 weeks
  Change from baseline to Week 4 in blood pressure
Change in Blod pressure | 12 weeks
  Change from baseline to Week 12 in blood pressure
Change in Heart rate | 4 weeks
  Change from baseline to Week 4 in heart rate
Change in Heart rate | 12 weeks
  Change from baseline to Week 12 in heart rate
Change in degree of vaginal atrophy | 12 weeks
  Change from baseline to Week 12 in the degree of vaginal atrophy. The assessment is made by okular gynocological examinations and graded mild, moderate and severe.
Urine infections | 12 weeks
  Number of urine infections during the study

CONTACTS AND LOCATIONS:
Overall Officials: Aino Fianu Jonasson, MD, PhD, Principal Investigator — Karolinska Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No